CLINICAL TRIAL: NCT02053545
Title: Haplo-identical Stem Cell Transplantation (SCT) for High-Risk Hematologic Malignancies With Post-Transplant In-Vivo T-cell Depletion
Brief Title: Haplo-identical SCT for High Risk (HR) Hematologic Malignancies w/Post-Transplant In-Vivo T-cell Depletion
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study closed with no enrollment.
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Reggie E Duerst, MD, Primary Investigator, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCT 0813 Haplo
Record Dates: First submitted 2013-12-31; First posted 2014-02-03 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Leukemia; Lymphoma; MDS
MeSH Terms: conditions — Leukemia; Lymphoma | interventions — Transplantation Conditioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Conditioning Regimen & GVHD Prophylaxis (Experimental): Stratum 1 (Refractory disease, relapse after previous transplant): Clofarabine, Melphalan,Thiotepa, Cyclophosphamide, Mesna, Tacrolimus and mycophenolate mofetil (MMF)
  Stratum 2 (Myeloid in remission): Busulfan, Fludarabine, Thiotepa, Cyclophosphamide, Mesna, Tacrolimus, MMF
  Stratum 3 (Lymphoid in remission): Fractionated total body irradiation (fTBI), Fludarabine, Thiotepa, Cyclophosphamide, Mesna, Tacrolimus, MMF
  Interventions: Drug: Conditioning Regimen & GVHD Prophylaxis

INTERVENTIONS:
Drug: Conditioning Regimen & GVHD Prophylaxis — Stratum 1 (Refractory disease, relapse after previous transplant): Radiation Therapy (if patient had prior Central Nervous System (CNS) disease), Clofarabine, Melphalan,Thiotepa, Stem Cell Transplant, Cyclophosphamide, Mesna, Tacrolimus and MMF
  Stratum 2 (Myeloid in remission): Radiation Therapy (if patient had prior CNS disease), Busulfan, Fludarabine, Thiotepa, Stem Cell Transplant, Cyclophosphamide, Mesna, Tacrolimus, MMF
  Stratum 3 (Lymphoid in remission): Radiation Therapy (if patient had prior CNS disease), TBI, Fludarabine, Thiotepa, Stem Cell Transplant, Cyclophosphamide, Mesna, Tacrolimus, MMF

SUMMARY:
Although a majority of children with leukemia and most hematological malignancies (Hodgkin's and Non-Hodgkin's lymphomas) can be cured with conventional chemotherapy, a subset of patients with resistant/recurrent high-risk disease are not cured with conventional treatment regimens. Investigators hypothesize that HSCT from a partially matched donor can be safe and effective for patients with very high risk hematologic malignancies when combined with post-transplant cyclophosphamide for prevention of graft-vs-host disease (GVHD).

DETAILED DESCRIPTION:
For patients whose disease cannot be brought into remission the prognoses are worse primarily due to high rates of post-HSCT relapse. For patients who have poor donor options (i.e., lack an adequately matched allogeneic marrow donor), the prognoses are worse for a successful outcome due to higher rates of treatment related mortality (TRM). Their options are to seek investigational treatments without HSCT or alternative investigational HSCT protocols for which they are eligible. Patients who have relapsed after an allogeneic HSCT are at high risk for either relapse or TRM after a subsequent HSCT, even if an additional state of complete remission can be achieved prior to the subsequent HSCT.

This current treatment protocol is designed to assess alternative HSCT treatments for patients with refractory/very high risk disease features and/or inadequate single sources of human leukocyte antigen (HLA)- matched -donor stem cells. The goal is to cure their hematological malignancy with the combination of chemotherapy and potentially destruction of cancerous cells by the new, donor immune cells.

For patients whose only potential for cure is allogeneic HSCT but who are lacking a well matched relative or unrelated donor source, haplo-identical donors (i.e., "half identical" donors) are a remaining option. However, without some form of immune manipulation of the donor marrow (e.g. pre-infusion in vitro or in the test tube/laboratory T-depletion, or depletion of donor T-cells), outcomes after haplo-identical HSCT have very poor results with unacceptable TRM, non-engraftment or severe graft-vs-host disease (GVHD)2 leading to fatal complications. GVHD is a complication that can occur after a stem cell or bone marrow transplant in which the newly transplanted donor cells attack the healthy tissues in the transplant recipient's body.

Thus, to better treat resistant leukemia, there is a need for either improved cytoreduction (pre-transplant reduction in the number of the cancer/leukemia cells) regimens for refractory disease, and/or for improved methods of eliminating cancer cells after the transplant has occurred.

Using well matched donors, investigators have studied the use of HSCT using mild chemotherapy but exploiting the donor cell immune reaction post-stem cell infusion to "allow" the reaction against leukemia and lymphoma cancer cells. This has generally proven ineffective for patients with disease not in remission at the time of transplant.

Thus new approaches to combat residual refractory disease are still needed. Also, for patients lacking well-matched donors, new methods to facilitate use of haplo-identical donors are needed.

Investigators hypothesize that HSCT from a partially matched (haplo-identical) related (usually sibling or parent or child) donor can be safe and effective for patients with very high risk hematologic malignancies when combined with an intensive, myeloablative (marrow destroying) cytoreduction treatment pre-HSCT followed by post-transplant cyclophosphamide for prevention of Graft Versus Host Disease (GVHD) in the recipient. This approach has been employed at other centers, primarily in adult recipients.2-4 One center's experience in pediatric patients demonstrated that non-relapse mortality was low and donor engraftment occurred in 12 of 12 patients.5 More experience with this approach is needed in pediatric HSCT patients.

In this Pilot Study, investigators hope to determine the likelihood that a myeloablative cytoreduction regimen followed by haplo-identical HSCT and high-dose post-transplant cyclophosphamide leads to adequate engraftment for high-risk hematologic malignancy patients. The patients that will be transplanted on this study are patients whose likelihood of survival without a transplant would be very low (<10-15 %, whether due to relapse after prior HSCT, poor disease control, or no matched donor available).

This treatment protocol does not involve an investigational drug but the combination of chemotherapy drugs in a new sequence/scheduling along with the use of haplo-identical donor stem cells. In this treatment protocol, patients will be treated in three different strata according to what defines their high-risk for a poor outcome. Each stratum will be comprised of a pre-transplant chemotherapy conditioning regimen followed by infusion of haplo-identical related donor marrow stem cells, followed in turn by post-transplant cyclophosphamide as immunosuppression to prophylax against GVHD.

The chemotherapeutic agents in this study, including cyclophosphamide, are routinely administered in children and adolescents for treatment. Cyclophosphamide is most commonly administered as a component of the pre-transplant cytoreduction therapy. However, for this treatment protocol investigators plan to assess the ability of utilizing a combined approach of the chemotherapeutic agents, with cyclophosphamide, as an effective prevention of GVHD infused after receiving a transplant from a closely matched (but not identical) family member.

The common elements of this research are high-dose cytoreduction therapy prior to HSCT, high-dose cyclophosphamide following HSCT and partially matched, related donor bone marrow cells as the source of stem cells infused for transplantation. The research question is the outcome of the patients treated with this combination. The cytoreduction regimen is tailored for the specific risk (prior HSCT, poor disease control vs no matched donor source of stem cells).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have confirmed diagnosis of hematologic malignancy (leukemia, lymphoma or MDS) with the following:
* Resistant/refractory hematologic malignancies (disease exceeding 5% of marrow cells by morphology, which is a description of white blood cell types as assessed via light microscopy; or with measurable extramedullary disease, which is detection of leukemia at sites other than blood and marrow. This includes disease that infiltrates into tissues other than the spleen and marrow. i.e. nodal disease, which is leukemia and/or lymphoma involving a lymph node or chloroma, which is a collection of leukemic cells forming a mass/tumor mass) (Stratum 1).
* Or have relapsed following an initial allogeneic HSCT (Stratum 1).
* And/or lack an adequately matched unrelated donor (URD) or unrelated cord blood (URB) hematopoietic stem cell (HSC) source (see protocol section 2) (Strata 1, 2 & 3).
* Adequate cardiac, pulmonary, renal, and hepatic functions
* Central vascular access providing a combined 3 access ports for all patients.
* Females of childbearing potential must have a negative pregnancy test prior to therapy. Pregnancy tests will only be done prior to therapy. Sexually active patients will be informed of the risk of not using adequate contraception.
* Recipient or legal guardian must be informed of the study, and have signed a consent form.
* Recipients must have a related haplo-identical donor.

Exclusion Criteria:

* High risk hematologic malignancies in remission (and no prior allogeneic HSCT), where allogeneic HSCT is indicated but an appropriately matched HSC source (sibling, unrelated adult or UCB) is available.
* Patients with systemic infections and/or organ dysfunction mandating a reduced intensity conditioning regimen are also excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2017-05-11 (Estimated); Study Completion 2017-05-11 (Actual)

PRIMARY OUTCOMES:
Cumulative non-relapse mortality at 100 days and 365 days post haplo-identical transplant | 1 Year
  Patients will be followed regularly for engraftment, complications, and disease control. Non-relapse mortality and overall survival will be recorded from date of HSCT.

SECONDARY OUTCOMES:
Cumulative acute and chronic GVHD, cumulative relapse rates, and overall survival and event free survival | 1 Year

OTHER OUTCOMES:
Engraftment Kinetics and Immune Reconstitution | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Reggie Duerst, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States